CLINICAL TRIAL: NCT04929080
Title: A Phase I/II Clinical Study of JS004, a Recombinant Humanized mAb Specific to B-and T-Lymphocyte Attenuator (BTLA), in Subjects With Head and Neck Cancer
Brief Title: The Safety and Efficacy of Multiple-dose of JS004 in Subject With HNC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS004-004
Record Dates: First submitted 2021-05-10; First posted 2021-06-18 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Head and Neck Squamous Cell Carcinom; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- JS004 200mg, Q3W until to 2 years (Experimental): Part A: phase I: 3-6; phase II: 66.
  Interventions: Biological: JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion
- JS004 600mg, Q3W until to 2 years (Experimental): Part A: phase I: 3-6; phase II: 66.
  Interventions: Biological: JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion
- 240mg JS001+100mg JS004, Q3W until to 2 years (Experimental): Part B: phase I: 6; phase II: 68.
  Interventions: Biological: JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion; Biological: JS001 and JS004
- 240mg JS001+200mg JS004, Q3W until to 2 years (Experimental): Part B: phase I: 6; phase II: 68.
  Interventions: Biological: JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion; Biological: JS001 and JS004

INTERVENTIONS:
Biological: JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion — 200mg:JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion
  Arms: 240mg JS001+100mg JS004, Q3W until to 2 years; 240mg JS001+200mg JS004, Q3W until to 2 years; JS004 200mg, Q3W until to 2 years
Biological: JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion — 600mg:JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion
  Arms: JS004 600mg, Q3W until to 2 years
Biological: JS001 and JS004 — Part B: 100mg JS004 + 240mg JS001 or 200mg JS004+ 240mg JS001
  Arms: 240mg JS001+100mg JS004, Q3W until to 2 years; 240mg JS001+200mg JS004, Q3W until to 2 years

SUMMARY:
A phase I/II clinical study of JS004 in subjects with head and neck cancer in China, to evaluate the safety, tolerability, PK, immunogenicity, antitumor activity and biomarkers of JS004, define the RP2D. A cycle is 21 days (3 weeks) which includes JS004 being administered IV Q3W and JS004 combine with JS001 being administered IV Q3W. All patients will be treated until disease progression per RECIST v1.1 and iRECIST, or intolerable toxicity per CTCAE 5.0, withdrawal of consent, or end of the study, whichever occurs first.Disease progression must be confirmed at least 4 weeks but no longer than 8 weeks after initial documentation of progression.

ELIGIBILITY:
Inclusion criteria:

1.Males and females ≥ 18 and ≤ 80 years of age; 2.Recurrent or metastatic squamous cell carcinoma of the head and neck and nasopharyngeal carcinoma confirmed histologically or cytologically are no longer suitable for local treatment such as surgery or radiotherapy； 3.Has received at least a first-line standard regimen for relapsed and metastatic disease and has progressed during or after treatment; 4.The Eastern Cooperative Oncology Group (ECOG) had a physical status score of 0 or 1. 5.Life expectancy ≥12 weeks; 6.At least one measurable lesion per RECISTv1.1 and iRECIST; 7.Willingness to provide consent for fresh pre-treatment biopsies, or,an archival specimen could be required within two years prior to the first dose of study drug; 8.Adequate organ and marrow function per protocol specifically defined; 9.Females of childbearing potential ,and males who are sexually active with a female partner of childbearing potential, must use effective contraception from time of screening, and must agree to continue using such precautions for 60 days after the final dose of JS004; 10.All acute toxic reactions caused by previous anti-tumor therapy, surgery or radiotherapy were alleviated to grade 0-1 (according to NCI-CTCAE version 5.0) or to the level specified by the inclusion/exclusion criteria.Except for hair loss, pigmentation, or other toxicity that the researcher believes does not pose a safety risk to the subject, and does not affect treatment compliance. 11.Able to understand and willing to sign the Informed Consent Form;

Exclusion criteria:

1.This is a histologically or cytologically confirmed salivary adenocarcinoma or other non-squamous cell carcinoma;nasopharyngeal carcinoma is not applicable. 2.Previously received anti-BTLA or anti-HVEM antibody treatment. 3.There are necrotic lesions, and the investigator has assessed the risk of hemorrhage 4.Other malignancies were diagnosed within 5 years prior to study entry; 5.There are uncontrolled or symptomatic active central nervous system (CNS) metastases; 6.Poor control of pleural effusion, peritoneal effusion, or pericardial effusion; 7.Peripheral neuropathy or hearing loss≥Grade 2 (according to NCI-CTCAE 5.0); 8.Pregnant or breastfeeding women.

9.Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; 10.Idiopathic pulmonary fibrosis, drug-induced pneumonia, mechanized pneumonia (i.e., bronchiolitis obliterans), radiation pneumonia with clinical symptoms or requiring steroid treatment, active pneumonia, or other moderate to severe lung diseases that seriously affect lung function. 11.The following conditions occurred within 6 months before the first study administration: myocardial infarction, severe/unstable angina pectoris, NYHA grade 2 or higher cardiac insufficiency, clinically significant supraventricular or ventricular arrhythmia, and symptomatic congestion Heart failure 12.Poorly controlled hypertension; hypertensive crisis or hypertensive encephalopathy occurred within 6 months of the first administration; 13. Those who are known to be allergic to the study drug or any of its excipients, or have severe allergic reactions to other monoclonal antibodies; 14. Have received the following drugs or treatments before the first study drug treatment:

1. Major surgery has been performed within 28 days before the first study administration.
2. Received systemic anti-tumor therapy within 28 days before the first study administration;
3. Participated in other intervention studies within 28 days before the first study dose;
4. Received systemic immunomodulatory drug treatment within 14 days before the first study administration or within 5 half-lives of the drug;
5. Received systemic corticosteroids or other systemic immunosuppressants within 14 days before the first study administration;
6. Received oral or intravenous antibiotic treatment within 14 days before the first study administration (except for the case of prophylactic use of antibiotics);
7. Any live vaccine has been vaccinated within 28 days before the first study administration; 15. Have a history of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, blood vessel thrombosis related to antiphospholipid syndrome Formation, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis or glomerulonephritis; 16. Severe infections (NCI-CTCAE> level 2) occurred within 28 days before the first study administration, such as severe pneumonia, bacteremia, and infectious comorbidities that require hospitalization.

17. Active infections, including tuberculosis (clinical diagnosis includes clinical history, physical examination and imaging findings, and TB examination according to local medical routines), hepatitis B, hepatitis C or human immunodeficiency virus (HIV antibody positive) ； 18. The presence of other serious physical or mental illnesses or abnormal laboratory tests, or alcoholism, drug abuse, etc., may increase the risk of participating in the study, affect treatment compliance, or interfere with the results of the study, and other cases determined by the investigator to be unsuitable for participation Patients in this study."

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events (AE) and serious adverse events (SAE) were assessed | 2 years
  Incidence and severity of adverse events (AE) and serious adverse events (SAE) as assessed according to NCI-CTCAE 5.0, as well as abnormalities in vital signs, electrocardiogram, and laboratory tests
ORR evaluated according to RECIST 1.1 | 2 years
  Objective Response Rate(ORR) evaluated according to RECIST 1.1

SECONDARY OUTCOMES:
Phase II Recommended Dose of JS004 (RP2D-A) and JS004 combined with JS001(RP2D-B) | 2 years
  Phase II Recommended Dose of JS004 (RP2D-A) and JS004 combined with JS001(RP2D-B)
DCR | 2 years
  Disease Control Rate (DCR)
ADA/Nab rate | 2 years
  the rate of Anti-drug body (ADA) and neutralizing antibody (Nab)
Cmax | 2 years
  Maximum Plasma Concentration(Cmax) after injection of JS004
DOR | 2 years
  Duration of Response
PFS | 2 years
  Progression-free survival evaluated according to RECIST 1.1
OS | 2 years
  Overall survival
6-month OS rate | 6 months
  6-month overall survival rate

OTHER OUTCOMES:
Predictive biomarkers | 2 years
  Predictive biomarkers, including but not limited to, BTLA and HVEM
Ctrough | 2 years
  trough Plasma Concentration (Ctrough) after injection of JS004
Tmax | 2 years
  Perk Time(Tmax) after injection of JS004
AUC | 2 years
  Area Under the Cure(AUC) after injection of JS004
t1/2 | 2 years
  t1/2 after injection of JS004
Plasma Clearence(CL) | 2 years
  Plasma Clearence(CL) after injection of JS004
volume of distribution of steady state(Vss) | 2 years
  volume of distribution of steady state(Vss) after multiple dose injection of JS004

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital, Chengdu, China